CLINICAL TRIAL: NCT07208058
Title: An Open-label, Single-arm, Multicenter, Phase III Clinical Study to Evaluate the Efficacy, Safety, and Tolerability of Plonmarlimab in Subjects With Relapsed/Refractory Rheumatic and Immunologic Disease-associated Haemophagocytic Lymphohistiocytosis (Also Known as Macrophage Activation Syndrome [MAS])
Brief Title: A Phase III Clinical Study to Evaluate the Efficacy, Safety, and Tolerability of Plonmarlimab in Subjects With Relapsed/Refractory Rheumatic and Immunologic Disease-associated Haemophagocytic Lymphohistiocytosis (Also Known as Macrophage Activation Syndrome [MAS])
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: TJ Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THZ0103-MAS301
Record Dates: First submitted 2025-09-27; First posted 2025-10-06 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Relapsed/Refractory Rheumatic and Immunologic Disease-associated Haemophagocytic Lymphohistiocytosis
MeSH Terms: conditions — Recurrence | interventions — plonmarlimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plonmarlimab (Experimental)
  Interventions: Drug: Plonmarlimab

INTERVENTIONS:
Drug: Plonmarlimab — Subjects will receive Plonmarlimab 10 mg/kg by intravenous injection once weekly from Week 1 to Week 3, and Plonmarlimab 6 mg/kg by intravenous injection once weekly from Week 4 to Week 8 (10 mg/kg QW×3 + 6 mg/kg QW×5).

SUMMARY:
A study designed to evaluate the efficacy, safety, immunogenicity, PK, and PD characteristics of Plonmarlimab in patients with relapsed/refractory rheumatic and immunologic disease-associated MAS, and to explore biomarkers related to the efficacy of Plonmarlimab.

ELIGIBILITY:
Inclusion Criteria:

* Age: 16 to 80 years (inclusive), of any gender.
* The subject is willing to participate in this study and voluntarily signs the informed consent form. For minor subjects aged 16 years (inclusive) to less than 18 years, written informed consent must be signed by both the subject and the subject's legal guardian.
* Diagnosed with a rheumatic and immunological disease.
* Diagnosed with haemophagocytic lymphohistiocytosis (HLH) according to the HLH-2004 diagnostic criteria (excluding molecular diagnosis)
* No response to/or dependence on/intolerance to/or worsening during high-dose corticosteroid therapy. High-dose corticosteroid therapy: at least 1.5-2.0 mg/kg/d of prednisone or its equivalent dose for 3 consecutive days, including methylprednisolone pulse therapy (15-30 mg/kg/d, maximum dose 1 g/d, for 3-5 days).

Exclusion Criteria:

* Confirmed or suspected primary haemophagocytic lymphohistiocytosis (pHLH).
* HLH induced by infection (including but not limited to EBV-HLH) or treatment (including but not limited to drugs such as CAR-T cells, TCEs, ADCs).
* History of other active neoplasm malignant within 5 years prior to screening, with the exception of successfully treated cutaneous basal cell or squamous cell carcinoma, or localised neoplasms that have been adequately treated with curative intent, including but not limited to, uterine carcinoma in situ, breast cancer in situ, thyroid cancer, etc.; asymptomatic, localised prostate cancer confirmed to have no metastasis and not requiring treatment, etc. Prior to receiving the investigational drug, an assessment by an oncology specialist is required to clarify the current status of the neoplasm malignant and to rule out the possibility of HLH secondary to the neoplasm malignant.
* History of allergy to any component of the investigational drug.
* Lung disorder: including but not limited to asthma, chronic obstructive pulmonary disease, interstitial lung disease, alveolar proteinosis, pulmonary granulomatosis, etc., and abnormal pulmonary function tests: forced vital capacity (FVC) <80% of predicted value, or FEV1/FVC <70%, etc.; or the investigator's comprehensive assessment concludes that the subject has a pre-existing lung disease that significantly affects pulmonary function and is unsuitable for participation in this clinical study.
* Cardiovascular disorder: history of acute myocardial infarction or unstable angina pectoris, severe arrhythmia (multifocal frequent premature ventricular contractions, ventricular tachycardia, ventricular fibrillation), etc., within the last 6 months; New York Heart Association (NYHA) functional class III-IV.
* Infection: Presence of an infection deemed uncontrollable by the investigator during the screening period [including but not limited to tuberculosis, active syphilis infection, viral infection (EBV, CMV, COVID-19, active hepatitis B, active hepatitis C, human immunodeficiency virus), other bacterial infections (including but not limited to atypical mycobacteria, Shigella, Salmonella, Campylobacter, etc.)].
* Abnormal renal function: creatinine (Cr) or urea/blood urea nitrogen (BUN) test value >1.5 times the upper limit of normal (ULN); or eGFR <60 mL/min during the screening period, calculated using the MDRD formula: eGFR [mL/(min × 1.73 m2)] = 186 × serum creatinine (mg/dL)-1.154 × age (years)-0.203 × (0.742 if female) × 1.233.
* Haematological diseases: Subjects with a past or current history of haematological diseases (including but not limited to, myelofibrosis, aplastic anaemia, leukaemia, lymphoma, etc.).
* Surgery or other conditions: Planned surgery or any other medical history, laboratory test abnormal, or other condition that, in the investigator's judgment, makes the subject unsuitable for participation in this study.
* Transplant: History of major organ transplant (e.g., heart, lung, kidney, liver) or haematopoietic stem cell/bone marrow transplant.
* Other diseases: Subject currently has a clinically significant and clinically unstable or inadequately controlled acute or chronic disease (e.g., acute pneumonia, pulmonary arterial hypertension, diabetic ketoacidosis, pancreatitis acute, etc.).
* Pregnant or lactating women.
* Participation in any clinical trial (including investigational vaccines) treatment or use of an invasive investigational medical device within 3 months prior to enrolment, or currently enrolled in an interventional study.
* Received live vaccine within 30 days prior to screening.
* Evidence of alcohol abuse within 3 months prior to screening or current abuse, identified through medical history inquiry.
* Other conditions that, in the investigator's opinion, make the subject unsuitable for participation in this clinical study. For example, any condition that may increase the risks associated with the subject's participation in the study, or may interfere with the evaluation of the investigational drug or confound the interpretation of the study results.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | at the end of Week 8

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Children's Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang